CLINICAL TRIAL: NCT05789303
Title: Phase II Study of Belantamab Mafodotin in Combination With Carfilzomib, Pomalidomide, and Dexamethasone (KPd) in Patients With Relapsed Multiple Myeloma
Brief Title: Study of Belantamab Mafodotin With Carfilzomib, Pomalidomide, and Dexamethasone in Relapsed Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-1781
Record Dates: First submitted 2023-03-23; First posted 2023-03-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Relapse Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; carfilzomib; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: No Prior CAR T-Cell Therapy (Experimental): This cohort will consist of 19 participants who have not had CAR T-Cell Therapy. Participants will receive belantamab mafodotin, carfilzomib, pomalidomide and dexamethasone.
  Interventions: Drug: Belantamab mafodotin; Drug: Carfilzomib; Drug: Pomalidomide; Drug: Dexamethasone
- Cohort 2: Prior CAR T-Cell Therapy (Experimental): This cohort will consist of 64 participants who have had prior CAR T-Cell Therapy. Participants will receive belantamab mafodotin, carfilzomib, pomalidomide and dexamethasone.
  Interventions: Drug: Belantamab mafodotin; Drug: Carfilzomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — Cycles 1, 3, 5, 7, etc. (odd numbered cycles): 1.9 mg/kg IV on Day 1 (28-day cycles)
  Other Names: Blenrep
Drug: Carfilzomib — Cycle 1: 20 mg/m2 on Day 1, then 56 mg/m2 on Days 8/15
  Cycles 2-8: 56 mg/m2 on Days 1/8/15
  Cycles 9+: 56 mg/m2 on Days 1/15
  Other Names: Kyprolis
Drug: Pomalidomide — 3 mg Day 1-21 of 28-day Cycle
  Other Names: Pomalyst
Drug: Dexamethasone — Cycles 1-4: 40 mg Days 1/8/15/22
  Cycles 5+: 20 mg Days 1/8/15/22

SUMMARY:
Doctors leading this study hope to learn if the combination of belantamab mafodotin, carfilzomib, pomalidomide, and dexamethasone is effective and safe when given to people who have multiple myeloma that has gotten worse and is not responding to standard drugs that are used for treating multiple myeloma, including chimeric antigen receptor T-cell therapy.

Participation in this research will last about 6 -24 months, but it may be less or more depending on your response to treatment.

DETAILED DESCRIPTION:
Doctors leading this study hope to learn if the combination of belantamab mafodotin, carfilzomib, pomalidomide, and dexamethasone is effective and safe when given to people who have multiple myeloma that has gotten worse and is not responding to standard drugs that are used for treating multiple myeloma, including chimeric antigen receptor T-cell therapy.

Participation in this research will last about 6 -24 months, but it may be less or more depending on your response to treatment.

The purpose of this research is to gather information on the safety and effectiveness of belantamab mafodotin, carfilzomib, pomalidomide, and dexamethasone for patients with a history of two or more prior lines of myeloma therapy. This combination is not FDA-approved, although carfilzomib and pomalidomide, are separately FDA-approved agents in combination with dexamethasone.

ELIGIBILITY:
1. Subject must be ≥ 18 years of age.
2. Life expectancy of more than three months.
3. Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
4. Subject must have adequate organ function, defined by clinically confirmed lab values set by the study team.
5. Female Subjects: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
6. Male Subjects: contraceptive should be used consistently with local regulations regarding the methods of contraception for those Subjects in clinical studies. Male Subjects are eligible to participate if they agree to the following during the intervention period and for six months after the last dose of study treatment to allow for clearance of any altered sperm:

   Refrain from donating sperm plus either:

   • Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

   OR

   • Must agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females).
7. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0) must be ≤ Grade 1 at the time of enrollment except for alopecia and Grade 2 peripheral neuropathy.
8. Subject must be able to understand the study procedures and agree to participate in the study by providing written informed consent.
9. Subject must be willing to comply with the requirements consistent with the belantamab mafodotin and pomalidomide Risk Evaluation and Mitigation Strategy (REMS) programs.

   DISEASE-RELATED:
10. Subjects with relapsed or refractory multiple myeloma requiring systemic therapy, who have progressed after 2+ prior lines of anti-myeloma treatments. A line of therapy consists of ≥1 complete cycle of a single agent, a regimen consisting of a combination of several drugs, or a planned sequential therapy of various regimens.
11. Subjects may be exposed to lenalidomide, bortezomib, daratumumab, elotuzumab, pomalidomide and/or carfilzomib.
12. If NO prior CAR T-cell therapy: Subjects who have been deemed refractory to EITHER carfilzomib or pomalidomide are permitted but subjects cannot be refractory to both carfilzomib and pomalidomide. Refractoriness is defined here as disease which was non-responsive or progressive while on therapy or within 60 days of the last treatment in patients who had achieved a minimal response or better on prior therapy.
13. If prior CAR T-cell therapy: Subjects whose most recent line of therapy was anti-B-cell maturation antigen (BCMA) targeted CAR T-cell therapy are permitted to enroll, regardless of carfilzomib/pomalidomide refractory status, if they meet criteria for progression.
14. Measurable disease, as indicated by one or more of the following:

    1. Serum M-protein of 0.5 g/dL of greater. If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement (i.e. M-spike in the beta region), then quantitative immunoglobulin levels are acceptable (Immunoglobulin-A, Immunoglobulin-M, or Immunoglobulin-D > 600 mg/dL or Immunoglobulin-G> 1100 mg/dL).
    2. Urine M-protein ≥ 200 mg/24 hours.
    3. Involved serum free light chains ≥ 10 mg/dL provided that free light chain ratio is abnormal.
15. Subjects must receive insurance approval for pomalidomide and dexamethasone.

Exclusion criteria

Disease Related

1. Waldenström's macroglobulinemia, systemic amyloidosis, POEMS syndrome, or plasma cell leukemia at the time of screening.
2. Radiotherapy to multiple sites within 3 weeks before start of protocol treatment (localized radiotherapy to a single site 1 week before start is permissible).
3. Subject must not have used an investigational drug or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days preceding the first dose of study drug.
4. Prior refractory status to belantamab mafodotin. Concurrent Conditions
5. Current corneal epithelial disease except mild changes in corneal epithelium and mild punctate keratopathy.
6. Subject must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria.
7. Subject must not have presence of active renal condition (infection, requirement for dialysis or any other condition that could affect Subject's safety). Subjects with isolated proteinuria resulting from multiple myeloma (MM) are eligible, provided they fulfil the inclusion criteria.
8. Subject must not use contact lenses while participating in this study unless instructed by an ophthalmologist.
9. Subject must not be simultaneously enrolled in any interventional clinical trial.
10. Subject must not have had major surgery ≤ 2 weeks prior to initiating study treatment.
11. Subject must not have any evidence of active mucosal or internal bleeding.
12. Significant neuropathy (Grades 3-4, or Grade 2 with pain) at the time of the first dose and/or within 14 days before enrollment.
13. Subject must not have evidence of cardiovascular risk including any of the following:

    1. Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block. Controlled atrial fibrillation is not an exclusion.
    2. History of myocardial infarction, acute coronary syndromes, coronary angioplasty, or stenting or bypass grafting within three (3) months of screening.
    3. Class III or IV heart failure as defined by the New York Heart Association functional classification system
    4. Uncontrolled hypertension.
14. Subject must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
15. Subject must not have an active infection requiring treatment.
16. Subject with HIV infection will be excluded unless certain T-cell count, viral load and clinical qualifications are met as confirmed by the study doctor

    Note: consideration must be given to anti-retroviral and prophylactic antimicrobials that may have a drug:drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant.
17. Patients with Hepatitis B will be excluded unless certain clinical criteria are met as confirmed by the study doctor.
18. Subject must not have positive hepatitis C antibody test result or positive hepatitis C Ribonucleic acid test result at screening or within 3 months prior to first dose of study treatment unless the subject can meet the following criteria:

(1) Hepatitis C Ribonucleic acid test is negative (2) Receives successful anti-viral treatment (typically 8 weeks) followed by a negative nucleocapsid ribonucleic acid test after a washout period of at least 4 weeks.

Note: Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C test is obtained.

19. Subject must not have invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Subjects with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction.

20. Subject must not have any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with Subject's safety, obtaining informed consent or compliance to the study procedures.

21. Subjects must not be pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Very Good Partial Response (No Prior CAR T-Cell Therapy Cohort) | 6-24 months
  No prior CAR T-cell therapy cohort: Rate of very good partial response (VGPR) or better after 6 cycles according to the 2016 International Myeloma Working Group (IMWG) Response Criteria by Independent Review Committee (IRC).
Rate of Overall Response (Prior CAR T-Cell Therapy Cohort) | 6-24 months
  Prior CAR T-cell therapy cohort: Rate of overall response (ORR) as determined by investigator assessment.

SECONDARY OUTCOMES:
Overall Response Rate | 6-24 months
  Overall response rate as determined by the 2016 International Myeloma Working Group (IMWG) Response Criteria by Independent Review Committee (IRC) and investigator assessment.
Minimal Residual Disease Negativity Rate | 6-24 months
  Minimal Residual Disease (MRD) negativity rate as assessed by next generation sequencing (limit of detection < 10-5).
Progression-Free Survival | 6-24 months
  Progression-free survival of participants as determined by investigator assessment.
Overall Survival Among Participants | 6-24 months
  Overall survival of participants as determined by investigator assessment.
Frequency and Severity of Adverse Events (AEs)/ Serious Adverse Events | 6-24 months
  Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by the Common Terminology Criteria for Adverse Events v5.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Derman, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF